CLINICAL TRIAL: NCT02170142
Title: The Major Goal of This Project is to Characterize the Structural and Functional Development of Cortical Plate and White Matter of the Human Neonatal Brain From the Equivalent 30 Gestational Weeks to 45 Gestational Weeks.
Brief Title: Characterization of the Functional and Structural Development of the Human Neonatal Brain From 30 Wks to 45 Wks ga
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCT02170142; R01MH092535 (NIH)
Record Dates: First submitted 2014-06-13; First posted 2014-06-23 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Human Development
Keywords: MRI; perinatal brain; development, neonates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment: All subjects studied are normal healthy neonates without a condition. MRI will be used to assess normal brain development.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — non-invasive MRI techniques (DTI) and (ASL) will be used to assess normal brain development. DTI is capable of invasively delineating macroscopic anatomic components with high contrast and revealing structures at the microscopic level. ASL is capable of measuring cerebral blood flow and cerebral metabolic rate of oxygen.
  Other Names: 3T Philips Achieva MRI

SUMMARY:
The major goal of this project is to characterize the structural and functional development of cortical plate and white matter of the human neonatal brain from the equivalent 30 gestational weeks to 45 gestational weeks. The project is sponsored by niH R01MH092535. Furthermore, it is related to the blue print project of transcriptome atlas (niH RC2MH089921) with at least 36 million funding also sponsored by niH.

Revealing detailed anatomy at different equivalent gestational ages of human neonatal brain not only aids in understanding this highly ordered process, but also provides clues to detect abnormalities caused by genetic or environmental factors. Cerebral vascular measurements offer important information on cerebral metabolism. However, either anatomical or functional studies of human brain development during this period are surprisingly scarce. Diffusion tensor imaging (DTi), a recently developed technology of magnetic resonance imaging (MRi), is capable of noninvasively delineating macroscopic anatomical components with high contrast and revealing structures at the microscopic level. Cerebral vascular quantification including cerebral blood flow (CBF) and cerebral metabolic rate of oxygen (CMRo2) can also be obtained through noninvasive MRi, specifically arterial spin labeling (aSL) and T2-relaxation under spin tagging (TRuST) MRi. in this proposed study, the structure and function of neonatal brain will be explored using noninvasive MRi technologies. 102 infants will be recruited and no sedation will be applied during MRi. The resultant database will provide reference standards for diagnostic radiology of premature newborns and reveal the vascular activities of these newborn brains. Specifically, three aims will be achieved:

1. To delineate the anatomical development of complex structure in the cerebral wall and white matter tracts of neonatal brains at different equivalent gestational ages.
2. To quantify the cerebral blood flow and metabolic rate of oxygen of neonatal brain.
3. To correlate the structural and functional measurements with the gene transcriptome results.

DETAILED DESCRIPTION:
102 normal infants with age of 30 gestational weeks to 45 gestational weeks will be recruited in partnership with Division of Perinatal-neonatal Medicine which consists of neonatologists and pediatricians providing services in Parkland Health and Hospital System (PHHS) and Children's Medical Center (CMC) at Dallas. among 102 normal infants, there are 17 subjects at each following subgroup, 30-31 gestational weeks, 32-33 gestational weeks, 34-35 gestational weeks, 36-38 gestational weeks, 39-42 gestational week and 43-45 gestational weeks. once these infants are identified, structural and functional MRi data will be acquired with Philips 3T located at Radiology of CMC. The sequence details are as follows: DTi: a single-shot echo-planar imaging (ePi) sequence with SenSe parallel imaging scheme (SenSitivity encoding, reduction factor [?]2.5) will be used. The imaging matrix will be 112x112 with a field of view of 168x168mm (nominal resolution of 1.5mm), which will be zero filled to 256x256. axial slices of 1.5mm thickness will be acquired parallel to the anterior-posterior commissure line (aC-PC). a total of 65 slices will cover the entire hemisphere and brainstem without gap. The diffusion weighting will be encoded along 30 independent orientations and b value will be 1000s/mm2. imaging time for each sequence will be 5 minutes and 30 seconds. To increase signal noise ratio (SnR), two repetitions will be performed, resulting in DTi imaging time 11 minutes.

T1/T2-weighted imaging: Co-registered T2 weighted image, using a spin echo sequence, will be acquired with the echo time 120ms. Repetition time (TR) will be 4,500ms. The imaging resolution will be same as that of DTi. Co-registered FLaiR (Fluid attenuated inversion Recovery) T1 weighted image will also be acquired with the same field of view as that in diffusion tensor imaging. The T1/T2 weighted imaging time will be 5 minutes.

Resting state fMRi: Time series of 240 volumes of BoLD (Blood-oxygenation-Level-Dependent) images will be acquired with a single-shot gradient-recalled T2* weighted ePi pulse sequence. The details of the sequence are as follows: TR [?] 1500 ms; flip angle [?] 90o; slice thickness[?]2.5mm; matrix [?] 68 x 68; FoV [?] 168 mm x 168 mm; voxel size[?]2.5x2.5x2.5mm.

aSL and TRuST: Pseudo-Continuous aSL (PCaSL) sequence combined with a phase-contrast sequence will be used to obtain voxel level CBF estimation in units of ml blood per 100 g of tissue per min (ml/100g/min). The PCaSL sequence will be: field of view [?] 168x168mm, matrix[?]84x84, slice thickness[?]2mm, 50 axial slices acquired with zero gap, voxel size[?]2x2x2mm, SenSe factor[?]2.5. The phase contrast MRi will be performed with the slice location perpendicular to the four major feeding arteries (left/right internal carotid and vertebral arteries) at the level of cervical spine 3 (C3). Baseline venous oxygenation (Yv) will be determined in the sagittal sinus using a recently developed T2-Relaxation-under-Spin-Tagging (TRuST) MRi technique. The imaging parameters will be: voxel size 3.44x3.44x5mm3, four different T2-weightings with Tes of 0ms, 40ms, 80ms and 160ms, duration 1 minutes and 12 seconds. The imaging slice will be positioned axially to intersect the superior sagittal sinus at the level of approximately 10mm above the sinus congruence.

Single voxel MRS: Single voxel proton MRS with short Te will be acquired. PReSS (Point ReSolved Spectroscopy) will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Normal infants of both genders
2. Any race or ethnicity
3. Inborn preterm delivered from 30-45 weeks gestation
4. Medically stable for transport i.e. requiring at most a nasal canula < 2 liters for respiratory support.

Exclusion Criteria:

1. Infants not delivered from 30-45 weeks gestation
2. Infants who may have a neurological event at birth
3. Presence of known or suspected congenital anomalies such as chromosomal anomalies
4. Major congenital heart disease or congenital infection
5. Substance abuse and any grade>1 of intraventricular hemorrhage (IVH) by cranial ultrasound
6. Presence of cystic periventricular leukomalacia (PVL) by cranial ultrasound

Ages: 30 Weeks to 45 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates in the neonatal intensive care unit at Parkland Hospital
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
To observe normal brain development in neonates using MR imaging. | neonates from 30 wg to 45 wg

CONTACTS AND LOCATIONS:
Overall Officials: Hao Huang, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

REFERENCES:
- [Background] Huang H, Jeon T, Sedmak G, Pletikos M, Vasung L, Xu X, Yarowsky P, Richards LJ, Kostovic I, Sestan N, Mori S. Coupling diffusion imaging with histological and gene expression analysis to examine the dynamics of cortical areas across the fetal period of human brain development. Cereb Cortex. 2013 Nov;23(11):2620-31. doi: 10.1093/cercor/bhs241. Epub 2012 Aug 28. PMID 22933464
- See also: The BrainSpan atlas is a foundational resource for studying transcriptional mechanisms involved in human brain development. — http://www.brainspan.org/